CLINICAL TRIAL: NCT02725905
Title: Weight Management Counseling in Medical Schools: A Randomized Controlled Trial
Brief Title: Weight Management Counseling in Medical Schools
Acronym: MSWEIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Brown University (Other); Creighton University (Other); Georgetown University (Other); Harvard School of Public Health (HSPH) (Other); Oregon Health and Science University (Other); University of Alabama at Birmingham (Other); University of Iowa (Other); University of Louisville (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Judith Ockene, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 6730; 1R01CA194787-01A1 (NIH)
Record Dates: First submitted 2016-03-03; First posted 2016-04-01 (Estimated); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Obesity
Keywords: Weight Management Counseling; Medical School Education
MeSH Terms: conditions — Obesity | interventions — MME

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multi-Modal Education (MME) (Experimental): 1) The MME is a three year multi-modal educational intervention including a series of interactive learning components and interventions focused on integrated weight management counseling. Prior to its launch, each component of the curriculum will be refined using a school participatory approach to help ensure feasibility and acceptability.
  Interventions: Behavioral: Multi-Modal Education (MME)
- Traditional Education (TE) (Active Comparator): 2) The TE arm of the study includes the school's current curriculum which may include topics related to the treatment of weight management and obesity.
  Interventions: Behavioral: Traditional Education (TE)

INTERVENTIONS:
Behavioral: Multi-Modal Education (MME) — The MME curriculum focuses on developing weight management counseling (WMC) skills through several components: 1) a web course focused on WMC knowledge and clinical skill competencies; 2) WMC role-play exercises for an opportunity to use an algorithm to practice patient-centered WMC; 3) personal weight management exercises to increase awareness of "Assist" activities (e.g. daily food monitoring using mobile apps, etc); 4) obesity bias assessments, video, and discussions to modify attitudes of implicit weight bias; 5) a formative web-based encounter to interact with and receive feedback from a standardized patient; and 6) an enhanced clerkship rotation focusing on providing learning to preceptors and allowing students to observe preceptors counseling patients who are overweight or obese.
  Other Names: MME
  Arms: Multi-Modal Education (MME)
Behavioral: Traditional Education (TE) — Current curriculum may consist of topics related to biology, population health, or counseling skills. TE also may include sporadic stand-alone lectures or small group discussions conducted separately or as a part of a patient interviewing or behavioral course.
  Other Names: TE
  Arms: Traditional Education (TE)

SUMMARY:
Eight U.S. medical schools will be participating in the study: Weight Management Counseling in Medical Schools, also known as MSWEIGHT. This is a five-year randomized controlled trial (RCT) designed to compare the efficacy of two approaches to learning weight management counseling: 1)traditional education (TE) and; 2) multi-modal educational intervention (MME).

The study aims are to refine and compare the efficacy of MME to TE on observed student weight management counseling skills measured through the primary outcome, the Objective Structured Clinical Examination (OSCE).

DETAILED DESCRIPTION:
Eight U.S. medical schools are matched and then randomized to one of two educational interventions, MME or TE.

Schools randomized to TE represent "usual care" and will continue the current curriculum. The MME arm will build upon the traditional usual curriculum at the medical school. The MME is a multi-modal educational intervention of a series of interactive learning components focused on integrated weight management counseling. This MME intervention for weight management counseling uses the 5As model based on the updated American Heart Association (AHA) /American College of Cardiology (ACC) /The Obesity Society (TOS) and updated NHLBI guidelines.

ELIGIBILITY:
Inclusion Criteria:

The medical school has:

* Interest in WMC medical education reform.
* Curricula resources (e.g. academic computing) to facilitate web-course training and a system to maintain student contact.
* The willingness and ability to incorporate all components of MSWEIGHT into the medical school curriculum, require or strongly encourage students to participate, and award credit for completion.
* The willingness and ability to offer the WMC OSCE for third year medical students upon completion of the Family or Internal Medicine clerkship rotation.

Exclusion Criteria: The medical school does not have:

* The ability to incorporate all components of MSWEIGHT into the medical school curriculum.
* The ability to offer the WMC OSCE for third year medical students upon completion of the Family or Internal Medicine clerkship rotation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3199 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Mean Score on Objective Structured Clinical Exam (OSCE); MME and TE students will be compared regarding the mean score. | Up to 2 years
  The primary outcome is the OSCE, the standard method for evaluating medical students' skill level at U.S. medical schools. The investigators will compare the efficacy of MME to TE on weight management counseling skills assessed among two separate 3rd year student classes (pre and post MSWeight implementation). MME and TE students will be compared regarding the mean score.

SECONDARY OUTCOMES:
Mean self-efficacy score on 5As will be calculated as the mean of student's self-reported skill level (1=not at all skilled through 4=very skilled) on 7 items regarding patient counseling skills. | Up to Three Years
  Perceived self-efficacy skill on 5As (Ask, Advise, Assess, Assist, Arrange) will be assessed longitudinally as 1st Year medical students and then again as 3rd Year medical students. The investigators will compare the difference in self-efficacy between MME and TE. Mean self-efficacy score on 5As will be calculated as the mean of student's self-reported skill level on 7 items about patient counseling skills.
Percentage of students reporting 3 = moderately skilled or 4 = very skilled will be calculated on 7 items regarding patient counseling skills. | Upto Three Years
  Perceived self-efficacy skill on 5As (Ask, Advise, Assess, Assist, Arrange) will be assessed longitudinally as 1st Year medical students and then again as 3rd Year medical students. The investigators will compare the percentage of students reporting moderately skilled to very skilled in patient counseling skills in MME and in TE. Percentage of students reporting on self-efficacy will be calculated on 7 items about patient counseling skills.

CONTACTS AND LOCATIONS:
Overall Officials: Judith K Ockene, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (8):
- United States (8):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Georgetown University School of Medicine, Washington D.C., District of Columbia
  - University of Iowa Carver College of Medicine, Iowa City, Iowa
  - University of Louisville School of Medicine, Louisville, Kentucky
  - Creighton University School of Medicine, Omaha, Nebraska
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania
  - Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No
The investigators plan to share data through the project website, publications, and presentations to key organizations. The plan is also to share the use of research tools, such as surveys, OSCE cases, and curricula materials, developed over the course of the study. At this time there is no plan to make individual participant data (IPD) available.

REFERENCES:
- [Background] Leblanc ES, O'Connor E, Whitlock EP, Patnode CD, Kapka T. Effectiveness of primary care-relevant treatments for obesity in adults: a systematic evidence review for the U.S. Preventive Services Task Force. Ann Intern Med. 2011 Oct 4;155(7):434-47. doi: 10.7326/0003-4819-155-7-201110040-00006. PMID 21969342
- [Background] Block JP, DeSalvo KB, Fisher WP. Are physicians equipped to address the obesity epidemic? Knowledge and attitudes of internal medicine residents. Prev Med. 2003 Jun;36(6):669-75. doi: 10.1016/s0091-7435(03)00055-0. PMID 12744909
- [Background] Vitolins MZ, Crandall S, Miller D, Ip E, Marion G, Spangler JG. Obesity educational interventions in U.S. medical schools: a systematic review and identified gaps. Teach Learn Med. 2012;24(3):267-72. doi: 10.1080/10401334.2012.692286. PMID 22775792
- [Background] Forman-Hoffman V, Little A, Wahls T. Barriers to obesity management: a pilot study of primary care clinicians. BMC Fam Pract. 2006 Jun 6;7:35. doi: 10.1186/1471-2296-7-35. PMID 16756673
- [Background] Kristeller JL, Hoerr RA. Physician attitudes toward managing obesity: differences among six specialty groups. Prev Med. 1997 Jul-Aug;26(4):542-9. doi: 10.1006/pmed.1997.0171. PMID 9245677
- [Background] Davis NJ, Shishodia H, Taqui B, Dumfeh C, Wylie-Rosett J. Resident physician attitudes and competence about obesity treatment: need for improved education. Med Educ Online. 2008 May 2;13:5. doi: 10.3885/meo.2008.Res00257. PMID 20165535
- [Background] Adams KM, Kohlmeier M, Zeisel SH. Nutrition education in U.S. medical schools: latest update of a national survey. Acad Med. 2010 Sep;85(9):1537-42. doi: 10.1097/ACM.0b013e3181eab71b. PMID 20736683
- [Background] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2985-3023. doi: 10.1016/j.jacc.2013.11.004. Epub 2013 Nov 12. No abstract available. PMID 24239920
- [Background] Chisholm A, Hart J, Mann KV, Harkness E, Peters S. Preparing medical students to facilitate lifestyle changes with obese patients: a systematic review of the literature. Acad Med. 2012 Jul;87(7):912-23. doi: 10.1097/ACM.0b013e3182580648. PMID 22622210